CLINICAL TRIAL: NCT02128334
Title: Prospective Multicenter Observational Program for Evaluation of Efficacy and Tolerability of the 6-month Depot Eligard 45 mg in Patients With Advanced Prostate Carcinoma in Routine Clinical Practice of Uro-Oncologists in the Russian Federation
Brief Title: An Observational Study Looking at How Well the Drug Eligard Works and How Well it is Tolerated by the Body of Patients With Advanced Prostate Carcinoma in the Russian Federation
Status: Completed | Type: Observational
Sponsor: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Other Study IDs: RU-EGD-NI-001
Record Dates: First submitted 2014-04-29; First posted 2014-05-01 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Advanced Prostate Carcinoma
Keywords: Uro-Oncologists; PSA; Eligard; prostate carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — luprolide acetate gel depot; Leuprolide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with advanced prostate carcinoma
  Interventions: Drug: Eligard 45 mg Exposure

INTERVENTIONS:
Drug: Eligard 45 mg Exposure — Subcutaneous injections
  Other Names: leuprorelin acetate

SUMMARY:
Eligard is a 6-month depot injection formulation that combines the active ingredient leuprorelin acetate (LA) with a biodegradable polymer matrix (Atrigel® delivery system). The 6-month (45 mg) formulation was approved for the Russian market in 2009. It has been shown to reduce testosterone and prostate-specific antigen (PSA) levels and to be well tolerated in several clinical trials. However, clinical trials are limited by strict patient inclusion and exclusion criteria. Therefore, the current non-interventional study aimed at investigating whether the efficacy and tolerability of the 6-month LA depot formulation could also be confirmed in a broad and heterogeneous patient population encountered in daily clinical practice in the Russian Federation.

This study will evaluate total serum PSA and testosterone levels, Quality of Life (QoL) of patients, demographic patient data, diagnosis and diagnostic findings in patients. It will provide analysis in different subgroups of patients depending on previous hormonal treatment and anamnesis of disease.

ELIGIBILITY:
Inclusion Criteria:

* All male patients > 18 years of age with advanced PCa to whom oncourologist decided to prescribe Eligard 45 mg

Exclusion Criteria:

* Patient participation in any clinical trials.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male patients >18 years of age with advanced prostate cancer (PCa) to whom Eligard 45 mg was prescribed
Sampling Method: Probability Sample
Enrollment: 645 (Actual)
Dates: Start 2013-09; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Percentage change in total serum PSA | Baseline and every 6 months until 24 months after treatment start
Percentage change in testosterone levels | Baseline and every 6 months until 24 months after treatment start

SECONDARY OUTCOMES:
Number of adverse drug reactions | Baseline to 24 months after treatment start
Mean change in QoL based on EuroQOL five dimensions questionnaire (EQ-5D) | Baseline to 24 months after treatment start

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Principal Investigator — Astellas Pharma Europe B.V.
Locations (52):
- Russia (52):
  - Site RU34 Private Practice, Abakan
  - Site RU23 Private Practice, Anapa
  - Site RU33 Private Practice, Belgorod
  - Site RU27 Private Practice, Irkutsk
  - Site RU29 Private Practice, Irkutsk
  - Site RU36 Private Practice, Izhevsk
  - Site RU60 Private Practice, Kostroma
  - Site RU10 Private Practice, Krasnodar
  - Site RU12 Private Practice, Krasnodar
  - Site RU13 Private Practice, Krasnodar
  - Site RU9 Private Practice, Krasnodar
  - Site RU35 Private Practice, Kursk
  - Site RU1 Private Practice, Moscow
  - Site RU11 Private Practice, Moscow
  - Site RU14 Private Practice, Moscow
  - Site RU15 Private Practice, Moscow
  - Site RU2 Private Practice, Moscow
  - Site RU20 Private Practice, Moscow
  - Site RU3 Private Practice, Moscow
  - Site RU32 Private Practice, Moscow
  - Site RU4 Private Practice, Moscow
  - Site RU42 Private Practice, Moscow
  - Site RU44 Private Practice, Moscow
  - Site RU55 Private Practice, Moscow
  - Site RU56 Private Practice, Moscow
  - Site RU6 Private Practice, Moscow
  - Site RU61 Private Practice, Moscow
  - Site RU7 Private Practice, Moscow
  - Site RU71 Private Practice, Moscow
  - Site RU72 Private Practice, Moscow
  - Site RU8 Private Practice, Moscow
  - Site RU21 Private Practice, Nizhny Novgorod
  - Site RU63 Private Practice, Nizhny Novgorod
  - Site RU64 Private Practice, Nizhny Novgorod
  - Site RU53 Private Practice, Novosibirsk
  - Site RU30 Private Practice, Omsk
  - Site RU18 Private Practice, Orenburg
  - Site RU66 Private Practice, Orenburg
  - Site RU68 Private Practice, Oryol
  - Site RU37 Private Practice, Petrozavodsk
  - Site RU40 Private Practice, Ryazan
  - Site RU73 Private Practice, Ryazan
  - Site RU17 Private Practice, Saint Petersburg
  - Site RU19 Private Practice, Saint Petersburg
  - Site RU65 Private Practice, Saint Petersburg
  - Site RU76 Private Practice, Saint Petersburg
  - Site RU59 Private Practice, Stavropol
  - Site RU25 Private Practice, Syktyvkar
  - Site RU54 Private Practice, Tver'
  - Site RU26 Private Practice, Yekaterinburg
  - Site RU43 Private Practice, Yekaterinburg
  - Site RU58 Private Practice, Yekaterinburg